CLINICAL TRIAL: NCT06993974
Title: Clinical Study to Evaluate Safety and Efficacy of Nitazoxanide in Patients With Ulcerative Colitis.
Brief Title: Nitazoxanide in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Prof. Dr. Ahmed Ibrahim Mohammed El Mallah, faculty of pharmacy, Alexandria University. (Unknown); Assoc. Prof. Dr. Noha Alaa Eldin Hassan Hamdy, Faculty of pharmacy, Alexandria University. (Unknown); Assoc. Prof. Dr. Ibrahim Fathi Amer, Faculty of Medecine, Kafr Elsheikh University. (Unknown)
Responsible Party: Principal Investigator, Reham ELshafeiy, Clinical pharmacist, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4444
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group, n =35: who will receive 1 g mesalamine three times daily for 3 months.
  Interventions: Drug: Mesalamine
- Nitazoxanide group (Active Comparator): Nitazoxanide group, n= 35: will receive 1 g mesalamine three times daily plus nitazoxanide 500 mg twice daily for 3 months.
  Interventions: Drug: Mesalamine; Drug: Nitazoxanide

INTERVENTIONS:
Drug: Mesalamine — Mesalamine or 5-amino salicylic acid (5-ASA), plays a crucial role in the treatment of ulcerative colitis (UC). It is the first-line therapy for mild to moderate cases of UC and is considered a cornerstone in its management.
Drug: Nitazoxanide — Nitazoxanide is an FDA-approved oral medication used to treat protozoal infections and is also effective against metronidazole-resistant Clostridium difficile colitis.
  Arms: Nitazoxanide group

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory bowel Disease (IBD) that primarily affects the rectum and colon. The severity and persistence of mucosal inflammation are associated with morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both male and female will be included
* Mild and moderate UC patients are already diagnosed and confirmed by endoscope and histopathology.

Exclusion Criteria:

* Breast feeding or pregnancy.
* Colorectal cancer patients.
* Patients with severe UC.
* Patients taking rectal or systemic steroids.
* Patients taking immunosuppressives or biological therapies.
* Addiction to alcohol and / or drugs.
* Known allergy to the studied medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
change in partial mayo score. | 3 months
  One non-invasive clinical measure for determining the severity of UC is the PMS. The composite score is derived from three subcategories: stool frequency, rectal bleeding, and physician's general assessment. The total score falls between 0 and 9

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt